CLINICAL TRIAL: NCT02231385
Title: Acetic Acid Colonoscopy Enhancement Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Nuovo Regina Margherita Hospital (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: The "ACE" Study
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer; Serrated Adenomas; Colon Nos Polypectomy Tubular Adenoma
Keywords: Colorectal cancer; Serrated adenomas; Screening; Adenoma detection rate; Polypectomy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Acetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetic Acid (Experimental): Subjects in Group A (study group) will undergo a standard colonoscopy. Once the right colon has been fully examined, acetic acid 2% will be sprayed and the right colon re-examined from cecum to hepatic flexure with within a frame-time of two minutes.
  Subjects in Group B (control group) will undergo a second examination of the right colon without acid acetic and within the same frame-time.
  Interventions: Drug: Acetic Acid
- Control Group (No Intervention): Subjects in Group A (study group) will undergo a standard colonoscopy. Once the right colon has been fully examined, acetic acid 2% will be sprayed and the right colon re-examined from cecum to hepatic flexure with within a frame-time of two minutes.
  Subjects in Group B (control group) will undergo a second examination of the right colon without acid acetic and within the same frame-time.

INTERVENTIONS:
Drug: Acetic Acid — Subjects in Group A (study group) will undergo a standard colonoscopy. Once the right colon has been fully examined, acetic acid 2% will be sprayed and the right colon re-examined from cecum to hepatic flexure with within a frame-time of two minutes.
  Subjects in Group B (control group) will undergo a second examination of the right colon without acid acetic and within the same frame-time.
  Arms: Acetic Acid

SUMMARY:
The purpose of this study is to compare the additional diagnostic yield obtained by using the acetic acid as vital substance to improve the detection of serrated lesions at colonoscopy.

Patients who are scheduled for screening, surveillance or diagnostic colonoscopy will be recruited to the study and randomized to one of two groups. Each enrolled subject will undergo two "back-to-back" procedures limited to the examination of the right colon.

Subjects in Group A (study group) will undergo a standard colonoscopy. Once the right colon has been fully examined, acetic acid 2% will be sprayed and the right colon re-examined from cecum to hepatic flexure with within a frame-time of two minutes. Subjects in Group B (control group) will undergo a second examination of the right colon without acid acetic and within the same frame-time.

Results from the two groups will be analyzed and compared, with primary outcome measures being detection rates for serrated lesions. Secondary outcome measures will include adenoma detection rate in the right colon or other locations, characteristics of polyps detected, including size and histological results.

Subjects will be followed through a 24-72 hour telephone interview for analysis of unexpected adverse events. Clinical results will be analyzed using various statistical measures of significance.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is >40 years old
2. The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Patients with a history of colonic resection;
2. Patients with inflammatory bowel disease;
3. Patients with a personal history of polyposis syndrome;
4. Patients with suspected chronic stricture potentially precluding complete colonoscopy;
5. Patients with diverticulitis or toxic megacolon;
6. Patients with a history of radiation therapy to abdomen or pelvis;
7. Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Additional serrated lesions diagnosed after acetic acid spraying | 12 months
  Primary outcome is the additional number of serrated lesions detected at the level of the right colon after spraying of acetic acid and compared with the number of the same lesions detected after a second examination of the right colon using standard white-light high definition scopes

SECONDARY OUTCOMES:
- Number of new adenoma detected at second right colon examination in both studies group | 12 months
Number of overall serrated and/or adenomatous lesions in the whole colon | 12 months
Characteristic of lesions detected (size, morphology) | 12 months
Complication rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan; Cesare Hassan, MD, Principal Investigator — Nuovo Regina Margherita Hospital
Locations (2):
- Italy (2):
  - Nuovo Regina Margherita Hospital, Rome
  - Humanitas Research Hospital, Rozzano, Milan